CLINICAL TRIAL: NCT04502797
Title: A Feasibility Study to Evaluate The Effect of the Electronic Patient Visit Assessment On Pain and Quality of Life for Patients With Head and Neck Cancer (HNC)
Acronym: ePVA
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19-01914
Record Dates: First submitted 2020-07-28; First posted 2020-08-06 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional: Electronic Patient Visit Assessment (ePVA) (Experimental): Participants diagnosed with head and neck cancer randomized to Electronic Patient Visit Assessment intervention
  Interventions: Behavioral: Electronic Patient Visit Assessment (ePVA)
- Usual care (No Intervention): Participants diagnosed with head and neck cancer randomized to usual care.

INTERVENTIONS:
Behavioral: Electronic Patient Visit Assessment (ePVA) — The ePVA is an mHealth clinical support tool. The ePVA consists of a patient-reported measure that focuses on symptoms common to HNC (i.e. pain, eye, ear, nasal, mouth, voice, fibrosis, edema, skin, gastrointestinal, fatigue, limitation in movement, sleep, breathing, difficulty eating or drinking, swallowing, communication, social activities, anxiety, depression, and daily activities). PROMIS® questionnaires (pain intensity 3a, fatigue 6a, sleep disturbance 6a, anxiety 6a, depression 6a) are embedded within the ePVA.
  Arms: Interventional: Electronic Patient Visit Assessment (ePVA)

SUMMARY:
This randomized, non-blinded, phase 0/I study will assess the feasibility of conducting a large randomized clinical trial to evaluate the efficacy of the ePVA to improve pain management and HRQoL in HNC. Thirty participants undergoing radiation therapy (RT) (with or without chemotherapy) will be randomized to: 1) ePVA intervention or 2) usual care. The intervention consists of participants completing the ePVA every other week during radiation therapy (RT), then weeks 4, 12, and 24 after end of RT. Automated reports of ePVA data, including pain reports and patient-reports of pain medications, will be sent to providers to inform their clinical decisions.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this study, an individual must meet all of the following criteria:

1. Histologically diagnosed HNC
2. Undergoing RT with or without chemotherapy,
3. English speaking,
4. aged 18 years or older.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Unable to attend scheduled appointment due to geographical, social or mental reseaons,
2. In the opinion of the investigator, is unable or unlikely to comply fully with the study requirements or procedures for any reason (e.g. cognitve or physical impairment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-10-08 (Actual); Primary Completion 2022-03-15 (Estimated); Study Completion 2022-03-15 (Estimated)

PRIMARY OUTCOMES:
Patient completion of 6 out of 7 assessments | 24 weeks
  This is defined as a binary yes/no variable as to whether a participant completed 6 out of 7 assessments.

SECONDARY OUTCOMES:
Change in health-related quality of life | Baseline, week 4, week 12, week 24
  Measured by EORTC QLQ-C30 global QoL/health scale, which consists of 30 questions, building five functional scales (physical, role, emotional, cognitive, social), a global QoL/health scale, symptom scales (fatigue, pain, nausea and vomiting, dyspnea, sleep disturbance, appetite loss, constipation and diarrhea) and perceived financial difficulties. The scale will be transformed to scores 0 to 100 (100 indicates best quality of life and 0 indicates least).
Change in pain severity | Baseline, Day 7, Day 21, Day 35
  Measured by European Organization for Research and Treatment of Cancer (EORTC) QLQ-H&N-35 pain scale. The scale will be transformed to scores 0 to 100 (0 indicates least and 100 indicates most symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Janet VanCleave, PhD, RN, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Rory Meyers College of Nursing, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to janet.vancleave@nyu.edu. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health.
Access Criteria: Requests may be directed to janet.vancleave@nyu.edu